CLINICAL TRIAL: NCT04440189
Title: Use of GID SVF-2 Device to Produce Autologous Adipose-Derived Stromal Vascular Fraction for Treatment of Osteoarthritis of the Knee: A Pivotal Medical Device Randomized Concurrent Controlled Study
Brief Title: Autologous Adipose-derived Stromal Vascular Fraction for Treatment of Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GID BIO, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GIDOA-03
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive an injection of Lactated Ringers in their index knee
  Interventions: Device: GID SVF-2 Device System
- Stromal Vascular Fraction (SVF) (Experimental): Subjects will receive an injection of Stromal Vascular Fraction in their index knee
  Interventions: Device: GID SVF-2 Device System

INTERVENTIONS:
Device: GID SVF-2 Device System — The GID SVF-2 Device System is used for harvesting, filtering, separating and concentrating autologous stromal vascular fraction from adipose tissue.

SUMMARY:
This is a pivotal study to evaluate the efficacy and safety of a single injection of autologous adipose-derived SVF produced using the GID SVF-2 device system for treatment of pain with concomitant improvement in function associated with osteoarthritis of the knee joint.

DETAILED DESCRIPTION:
This is a prospective, randomized, placebo controlled, parallel groups, double blind, multi-center, interventional study of subjects with osteoarthritis of the knee. Subjects will be randomized to receive an injection of LR (placebo) or SVF derived from their own adipose tissue (experimental).

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral or unilateral knee osteoarthritis as diagnosed on pre-op MRI using the Outerbridge Cartilage Classification as Grade II, Grade III, or Grade IV with full thickness lesion of the articular cartilage is less than 4.0 cm in any direction
2. Kellgren and Lawrence score grade 2-4 as diagnosed on X-Ray
3. Index knee must present with a score ≥8 using the WOMAC pain scale (A1 subscale, 20 total points)
4. Study Subjects must be willing to voluntarily give written Informed Consent to participate in the study and sign the Health Insurance Portability and Accountability Act (HIPAA) authorization before any study procedures are performed
5. Males and females 35-85 years old
6. Subjects with BMI ≥22 and ≤ 37
7. Subjects must speak, read and understand English
8. Subjects must be able to return for multiple follow-up visits
9. Subjects must have failed at least two conservative therapies for treatment of knee OA within the last 24 months (2 years), with one or more of the failed conservative therapies being from a-f:

   1. Physical Therapy: 6 week course of treatment
   2. Exercise Therapy: 6 week course of treatment
   3. Viscosupplementation injection in the knee for OA pain
   4. Steroid injection in the knee for OA pain
   5. Platelet-Rich Plasma (PRP) injection in the knee for OA pain
   6. Arthroscopic surgery including microfracture and/or debridement
   7. Braces or other support devices: therapy tried for at least 2 weeks
   8. Over the Counter (OTC) pain medication including NSAIDS, Acetaminophen, ASA: therapy tried for at least 2 weeks
   9. Prescription pain medication: therapy tried for at least 1 weeks
   10. Modification of Activities of Daily Living (ADL): therapy tried for at least 2 weeks
   11. Topical applications to the knee for OA pain: therapy tried for at least 2 weeks
   12. Supplements including glucosamine sulfate and chondroitin sulfate: therapy tried for at least 4 weeks
   13. Ice/Heat regimen: therapy tried for at least 2 weeks

Exclusion Criteria:

1. Subjects whose knee pain is caused by:

   i. unstable meniscal root tears or locked bucket handle meniscal tears ii. displaced meniscus tear iii. osteo chondritis dissecans iv. parameniscal, Baker's, or ganglion cysts v. lipoma arborescens vi. Hoffa's Pad Syndrome vii. acute ligament tears viii. diffuse edema ix. patellar mal-tracking or patellar dislocations
2. Outerbridge Scale Grade 0-I as diagnosed on MRI
3. Outerbridge Scale Grade IV where the full thickness lesion of the articular cartilage is greater than 4.0 cm in any direction, as diagnosed on MRI
4. Subjects with malignant neoplasms of the bone, cartilage, synovium or vasculature.
5. Subjects who have had surgery of either knee within 6 months prior to the surgery visit
6. Subjects who have had a major injury to either knee within 12 months prior to the surgery visit
7. Subjects who have had an injection into the intraarticular space of either knee in the prior 6 months, including corticosteroids, viscosupplementation, stromal vascular fraction (SVF), bone marrow stem cells, or platelet rich plasma
8. Subjects who have a diagnosis of gout with a flare in the past 12 months.
9. Subjects who have a diagnosis of Pes Anserine Bursitis with an event in the past 12 months.
10. Subjects who have had a diagnosed infection in the knee joint in the past 12 months.
11. Subject who have received a diagnosis of the following at any time: rheumatoid arthritis, lupus arthropathy, psoriatic arthritis, avascular necrosis, fibromyalgia, or neurogenic or vascular claudication
12. Diagnosis of severe bone deformity defined as greater than 10 degrees of either varus or valgus deformity
13. Subjects that are unwilling to stop taking prescription or over the counter pain medication 7 days prior to any visit (except Day 2 Post Treatment Visit).
14. Subjects that are allergic to lidocaine, epinephrine or valium
15. Subjects with a history of bleeding disorders, anticoagulation therapy that cannot be stopped as follows prior to injection; thrombolytics and anti-platelet medication including but not limited to Coumadin (warfarin) for 3 days, Plavix (colpidogrel) for 3 days, ASA/NSAIDs/fish oil supplements for 7 days, Xarelto® (rivaroxaban) for 24 hours
16. Subjects with systemic immunosuppressant use within 6 weeks from screening
17. Subjects with HIV or viral hepatitis
18. Subjects who have ever received a diagnosis of:

    chondrocalcinosis, Paget's disease or Villonodular synovitis
19. Subjects that use any form of tobacco, including e-cigarettes, more than once a week over the most recent 1 year period
20. Women that are pregnant or planning to become pregnant during the study
21. Subjects on long term oral steroids defined as longer than a 2-week taper.
22. History of any chemotherapy or radiation therapy on either leg or adipose harvest site
23. Subjects currently on workers' compensation

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index | 12 months
  The WOMAC is a self-administered questionnaire consisting of 14 items divided into 3 subscales, pain, stiffness and function. The primary efficacy will be achieved if the SVF dose group is shown to have a clinically meaningful improvement in pain and function at 12 months post-treatment, using the percent change in WOMAC score from baseline as the primary variable. The overall WOMAC score is normalized to a range of 0 to 100 points with a lower score indicating less symptoms of osteoarthritis.

SECONDARY OUTCOMES:
Adverse Events | 12 months
  Summary of device, treatment and procedure related adverse event rates and severity

CONTACTS AND LOCATIONS:
Overall Officials: William Cimino, PhD, Study Chair — GID BIO
Locations (9):
- United States (9):
  - UC Davis, Sacramento, California
  - Advanced Research LLC, Coral Springs, Florida
  - Tulane University, New Orleans, Louisiana
  - New Jersey Regenerative Institute, Cedar Knolls, New Jersey
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Jameson Crane Sports Medicine Institute, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Center for Cell Therapy and Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garza JR, Campbell RE, Tjoumakaris FP, Freedman KB, Miller LS, Santa Maria D, Tucker BS. Clinical Efficacy of Intra-articular Mesenchymal Stromal Cells for the Treatment of Knee Osteoarthritis: A Double-Blinded Prospective Randomized Controlled Clinical Trial. Am J Sports Med. 2020 Mar;48(3):588-598. doi: 10.1177/0363546519899923. PMID 32109160